CLINICAL TRIAL: NCT02520440
Title: Clinical Evaluation of Gastro Intestinal Failure, Multiple Organ Failure and Levels of Citrulline in Critical Ill Patients
Brief Title: INtestinal Failure, multiPle Organ Failure ANd CItrulline Assessment
Acronym: IN-PANCIA
Status: Completed | Type: Observational
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Dr. Nazzareno Fagoni, MD, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: NP 1769/2014
Record Dates: First submitted 2015-08-06; First posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Citrulline; Organ Failure, Multiple; Gastro Intestinal Failure; Intra Abdominal Pressure
Keywords: Citrulline; GIF; MOF; Calprotectina; intraabdominal pressure
MeSH Terms: conditions — Multiple Organ Failure | interventions — Glutamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GIF and/or MOF patients: Development during the ICU stay of gastro-intestinal failure and/or multiple organ failure. Investigators performed in each patient monitoring of plasmatic levels of Citrulline, monitoring of plasmatic levels of Arginine and Glutamine, and intra-abdominal pressure monitoring.
  Interventions: Biological: Monitoring of plasmatic levels of Citrulline; Device: Intra-abdominal pressure monitoring; Biological: Monitoring of plasmatic levels of Arginine and Glutamine
- Controls: patients admitted to ICU without gastrointestinal failure and/or multiple organ failure during the intensive care unit stay. Investigators performed in each patient monitoring of plasmatic levels of Citrulline, monitoring of plasmatic levels of Arginine and Glutamine, and intra-abdominal pressure monitoring.
  Interventions: Biological: Monitoring of plasmatic levels of Citrulline; Device: Intra-abdominal pressure monitoring; Biological: Monitoring of plasmatic levels of Arginine and Glutamine

INTERVENTIONS:
Biological: Monitoring of plasmatic levels of Citrulline — Measured plasma amino-acids levels
Device: Intra-abdominal pressure monitoring — Intra-abdominal Hypertension is defined as an average pressure of the day ≥ 12 mmHg; abdominal compartment syndrome is defined as a sustained (minimally two standardized measurements, performed 1-6 h apart) increase in Intra-abdominal pressure above 20 mmHg with new onset organ failure.
Biological: Monitoring of plasmatic levels of Arginine and Glutamine — Measured plasma amino-acids levels

SUMMARY:
The gastrointestinal dysfunction occurs frequently during the intensive care unit (ICU) stay and is associated with a worse prognosis.

The gastrointestinal failure (GIF) is diagnosed based on symptoms such as bowel distension, ileus, diarrhea, digestive bleeding, or intestinal ischemia. A GIF score based on has been demonstrated to be correlated with outcome, with higher scores indicating higher risk of death. However, GIF may be occult or clinical signs can go undetected in critically ill patients due to the frequent use of analgesic, sedative or neuromuscular blocking agents, acute neurologic diseases, or delirium.

Citrulline is a potential biomarker for small bowel function in critically ill patients with maintained renal function. Normal plasma citrulline levels (12-55 µmol/L) are determined by the balance between gut synthesis and kidney degradation.

GIF is involved in the pathogenesis of multiple organ dysfunctions and failures (MOF) through various mechanisms, and it is often associated with high intra-abdominal pressure (IAP). IAP greater than 12 mmHg, may lead to abdominal compartment syndrome (ACS) and MOF, including cardiac, respiratory and kidney failure. Studies have suggested that GIF can be the consequence rather than the cause of MOF.

The aim of this study is to investigate if plasma citrulline levels is associated with a clinical diagnosis of GIF, and may predict the development of MOF.

ELIGIBILITY:
Inclusion Criteria:

- Intensive Care Unit stay of at least 48 hours

Exclusion Criteria:

* Intensive Care Unit stay less than 48 hours
* abdominal trauma or surgery in the last 6 weeks
* inflammatory bowel disease
* a body mass index (BMI) ≥35
* terminal condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in ICU
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Development of Gastro Intestinal Failure, defined as the presence of three or more gastro-intestinal symptoms; and Multiple Organ Failure measured by SOFA score | within the first 30 days after admission in intensive care unit
  to investigate if plasma citrulline levels are associated with a clinical diagnosis of Gastro Intestinal Failure, and may predict the development of Multiple Organ Failure. Gastrointestinal Failure is defined as the presence of three or more coincident GI symptoms (igh gastric residual volumes (GRV) = maximum GRV above 500 ml at least once. Absent bowel sounds (BS) = BS not heard on careful auscultation. Vomiting/Regurgitation= visible vomiting or regurgitation in any amount. Diarrhoea = loose of liquid stool three or more times per day. Bowel distension= suspected or radiologically confirmed bowel dilatation in any bowel segment. GI bleeding= visible appearance of blood in vomit, nasogastric aspirate or stool.). MOF was defined as the failure of two or more organs or system according to the Sequential Organ Failure Assessment (SOFA)

SECONDARY OUTCOMES:
Correlation between intra abdominal hypertension (defined as an average of intra-abdominal pressure of the day ≥ 12 mmHg), and development of Gastro Intestinal Failure and Multiple Organ Failure | within the first 30 days after admission in intensive care unit
  to investigate if increasing of intra abdominal pressure is associated with a clinical diagnosis of Gastro Intestinal Failure, and may predict the development of Multiple Organ Failure. Intra-abdominal Hypertension (IAH) is defined as an average IAP of the day ≥ 12 mmHg; abdominal compartment syndrome (ACS) is defined as a sustained (minimally two standardized measurements, performed 1-6 h apart) increase in IAP above 20 mmHg with new onset organ failure.
Correlation between levels of Arginine and Glutamine in patients with Gastro Intestinal Failure and Multiple Organ Failure | within the first 30 days after admission in intensive care unit
  to investigate if plasma Arginine and Glutamine levels are associated with a clinical diagnosis of Gastro Intestinal Failure, and may predict the development of Multiple Organ Failure.

CONTACTS AND LOCATIONS:
Overall Officials: Nazzareno Fagoni, MD, Principal Investigator — Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia

REFERENCES:
- [Background] Carlson GL, Dark P. Acute intestinal failure. Curr Opin Crit Care. 2010 Aug;16(4):347-52. doi: 10.1097/MCC.0b013e328339fabe. PMID 20489609
- [Background] Piton G, Manzon C, Cypriani B, Carbonnel F, Capellier G. Acute intestinal failure in critically ill patients: is plasma citrulline the right marker? Intensive Care Med. 2011 Jun;37(6):911-7. doi: 10.1007/s00134-011-2172-x. Epub 2011 Mar 12. PMID 21400011
- [Background] Reintam A, Parm P, Kitus R, Starkopf J, Kern H. Gastrointestinal failure score in critically ill patients: a prospective observational study. Crit Care. 2008;12(4):R90. doi: 10.1186/cc6958. Epub 2008 Jul 14. PMID 18625051
- [Background] Malbrain ML, Cheatham ML, Kirkpatrick A, Sugrue M, Parr M, De Waele J, Balogh Z, Leppaniemi A, Olvera C, Ivatury R, D'Amours S, Wendon J, Hillman K, Johansson K, Kolkman K, Wilmer A. Results from the International Conference of Experts on Intra-abdominal Hypertension and Abdominal Compartment Syndrome. I. Definitions. Intensive Care Med. 2006 Nov;32(11):1722-32. doi: 10.1007/s00134-006-0349-5. Epub 2006 Sep 12. PMID 16967294
- [Background] Puleo F, Arvanitakis M, Van Gossum A, Preiser JC. Gut failure in the ICU. Semin Respir Crit Care Med. 2011 Oct;32(5):626-38. doi: 10.1055/s-0031-1287871. Epub 2011 Oct 11. PMID 21989698
- [Background] Piton G, Manzon C, Monnet E, Cypriani B, Barbot O, Navellou JC, Carbonnel F, Capellier G. Plasma citrulline kinetics and prognostic value in critically ill patients. Intensive Care Med. 2010 Apr;36(4):702-6. doi: 10.1007/s00134-010-1751-6. PMID 20084502